CLINICAL TRIAL: NCT01698463
Title: Tailored Exercise for Fall and Fracture Prevention in Older Adults: A Family Health Team Approach
Brief Title: Prescribe Exercise for Prevention of Falls and Fractures: A Family Health Team Approach
Acronym: PEPTEAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: The Centre for Family Medicine, Ontario (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 17664
Record Dates: First submitted 2012-08-30; First posted 2012-10-03 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2017-11

CONDITIONS: Fall and Fractures Prevention
Keywords: Falls, Fractures, Osteoporosis, Frailty, Older Adults.
MeSH Terms: conditions — Fractures, Bone; Osteoporosis; Frailty | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Identify Patients at Risk/Exercise Prescription (Other): The intervention was delivered in two visits and two follow-up phone calls. Physician identifies that the patient is at risk of falls or fractures Visit one: individualized exercise prescription by a physiotherapist. Visit two: motivational interviewing (behavioural counselling) by kinesiologist Phone call 1 and 2: Kinesiologist reviews behavioural components (action planning, coping planning, coping self-efficacy, intentions.
  Interventions: Other: Identification of patients at risk, tailored exercise prescription, motivational interviewing, review of behavioural outcomes

INTERVENTIONS:
Other: Identification of patients at risk, tailored exercise prescription, motivational interviewing, review of behavioural outcomes — The intervention was delivered in two visits and two follow-up phone calls.
  * Physician identifies that the patient is at risk of falls or fractures
  * Visit one: individualized exercise prescription by a physiotherapist.
  * Visit two: motivational interviewing (behavioural counselling) by kinesiologist
  * Phone call 1 and 2: Kinesiologist reviews behavioural components (action planning, coping planning, coping self-efficacy, intentions.

SUMMARY:
Falls and fractures are a leading cause of death and disability in the older adult population. The consequences of falls and fractures contribute substantially to health care costs and can have a significant negative impact on the quality of life of the individual. Exercise has been studied as an option to reduce fracture risk and prevent falls though improving balance and muscle strength. The prevention of falls is important, as a history of falls is strongly predictive of suffering another. Those who are at a high risk of fracture or falling require a patient specific assessment and individualized exercise prescription that is tailored to their needs. This kind of program may not be typically available within the community and at a low cost. These individuals may experience difficulty when trying to engage in exercise due to barriers such as a lack of transportation, and a lack of knowledge. As the first point of contact with the health care system for many family doctors are in the ideal position to deliver exercise advice to their patients. However, a lack of time and specialized skills in prescribing exercise make this difficult for many of them. As a result, family health teams who provide interdisciplinary patient centered care are becoming popular. In this model the care is shared and provided by the most appropriate team member (e.g. doctor, nurse, exercise specialist). Additionally, many exercise interventions do not include a behavior change aspect, which may be an important component when trying to get individuals to engage in a new health behavior like exercise. Therefore the purpose of this project is to assess the feasibility of implementing a tailored exercise program to those at high risk of falls or fractures over the age of 65 in a primary care setting using an interdisciplinary model of care that is based on a health behaviour change model.

DETAILED DESCRIPTION:
Falls and fractures together represent one of the leading causes of morbidity and mortality within the older adult population. Additionally, the consequences of falls and fractures contribute substantial costs to the health care system and negatively impact the quality of life of the individual. Given that Canada's aging population in increasing at an unprecedented rate, it is imperative that the prevention and management of falls and fractures is made a priority. One such population particularly vulnerable to falls and fractures are those diagnosed with osteoporosis or low bone mass.

It has been estimated that approximately 10 billion individuals have been diagnosed with osteoporosis and another 34 million are at risk with low bone mass. Osteoporosis-related fragility fractures are a common consequence of osteoporosis and result in increased morbidity and mortality. Approximately 50% of those who suffer a hip fracture do not regain their previous level of mobility and functional independence thus resulting in many of these individuals relying on the use of assistive devices.

Currently the emphasis of osteoporosis treatment and management is to prevent the occurrence of fragility fractures and the subsequent side effects that accompany them. A recent meta-analysis has shown that exercise can assist in the prevention and maintenance of bone loss in postmenopausal women. Other benefits of exercise such as increases in muscle strength and balance have been strongly established to indirectly prevent fractures through a reduction in falls risk. Those who are at a high risk of falls or fracture require patient specific assessment and individualized prescription that is not typically available within the community or at a low cost. Further, it may be difficult to engage these individuals if they have spent most of their life in a sedentary state and experience barriers such as a lack of transportation, and a lack of knowledge on appropriate types of exercise or how to initiate exercise into their daily living. Furthermore, many exercises may not be appropriate for all individuals depending on location of fracture and level of physical function. It has been emphasized that the focus should be on an individualized exercise program, which would encompass individual needs while recognizing individual limitations.

Family physicians may be in an ideal position to deliver an exercise prescription to a patient, as they are often the first point of contact with the health care system. However, there have been a number of problems cited with using family physicians to implement the delivery of an exercise prescription. Among those barriers, a lack of time and a lack of knowledge have been identified as the most problematic. An interdisciplinary family health team model of care is becoming increasingly important in regards to the treatment of chronic conditions such as osteoporosis. Family health teams provide an ideal form of care where team members work together to deliver the program and enhance adherence.

A limitation of many exercise interventions is that they fail to include a behavior change component which may be an important factor to consider when attempting to facilitate adherence to an exercise program. The Health Action Process Approach is a model of behavior change that has been widely used in a variety of health contexts including but not limited to physical activity. The rationale for the selection of this model is that it incorporates key principles of other behavior change models. Furthermore, the model has been cited as being a valid and reliable tool for predicting physical activity levels in older adults.

This project outlines an exercise intervention that is multidisciplinary in nature and tailored to the individual to be employed within an interdisciplinary family health team. Additionally, a behavior change component is built into this intervention with key principles such as action planning and coping planning that are based on the HAPA model to facilitate the uptake of physical activity in this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* > age 65
* Patient of the Centre for Family Medicine Family Health Team (CFFM FHT)

Have at least one of the following:

* 2 or more falls in the past 12 months
* age 75 +
* high risk of fracture based on the CAROC
* difficulty with walking or balance as determined by attending physician
* acute fall
* history of a fragility fracture after the age of 50

Exclusion Criteria:

* moderate to severe cognitive impairment
* moderate to severe neurologic impairment
* not able to communicate in English
* contraindications to exercise as determined by physician
* uncontrolled hypertension
* palliative care, current cancer, on dialysis
* participation in a similar exercise program including resistance training at least 3 times a week

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lora M Giangregorio, PhD, Principal Investigator — University of Waterloo
Locations (1):
- Centre for Family Medicine (CFFM), Kitchener, Ontario, Canada

REFERENCES:
- [Background] Boonen S, Dejaeger E, Vanderschueren D, Venken K, Bogaerts A, Verschueren S, Milisen K. Osteoporosis and osteoporotic fracture occurrence and prevention in the elderly: a geriatric perspective. Best Pract Res Clin Endocrinol Metab. 2008 Oct;22(5):765-85. doi: 10.1016/j.beem.2008.07.002. PMID 19028356
- [Background] Guideline for the prevention of falls in older persons. American Geriatrics Society, British Geriatrics Society, and American Academy of Orthopaedic Surgeons Panel on Falls Prevention. J Am Geriatr Soc. 2001 May;49(5):664-72. No abstract available. PMID 11380764
- [Background] Leslie WD, O'Donnell S, Jean S, Lagace C, Walsh P, Bancej C, Morin S, Hanley DA, Papaioannou A; Osteoporosis Surveillance Expert Working Group. Trends in hip fracture rates in Canada. JAMA. 2009 Aug 26;302(8):883-9. doi: 10.1001/jama.2009.1231. PMID 19706862
- [Background] Brown AP. Reducing falls in elderly people: A review of exercise interventions. Physiother Theory Pract 1999;15:59-68.
- [Background] Statistics Canada. Estimates of population, by age group and sex for July 1, Canada, provinces and territories, annual (CANSIM Table 051-0001). Ottawa: Statistics Canada 2010.
- [Background] World Health Organization. WHO Global Report on Falls Prevention in Older Age. Geneva, Switzerland: World Health Organization. 2007; Available at: http://www.who.int/ageing/publications/Falls_ prevention7March.pdf. Accessed Retrieved Aug, 2011.
- [Background] Consensus development conference: diagnosis, prophylaxis, and treatment of osteoporosis. Am J Med. 1993 Jun;94(6):646-50. doi: 10.1016/0002-9343(93)90218-e. No abstract available. PMID 8506892
- [Background] National Osteoporosis Foundation. America's bone health: the state of osteoporosis and low bone mass in our nation. Washington DC: National Osteoporosis Foundation. 2002.
- [Background] Ioannidis G, Papaioannou A, Hopman WM, Akhtar-Danesh N, Anastassiades T, Pickard L, Kennedy CC, Prior JC, Olszynski WP, Davison KS, Goltzman D, Thabane L, Gafni A, Papadimitropoulos EA, Brown JP, Josse RG, Hanley DA, Adachi JD. Relation between fractures and mortality: results from the Canadian Multicentre Osteoporosis Study. CMAJ. 2009 Sep 1;181(5):265-71. doi: 10.1503/cmaj.081720. Epub 2009 Aug 4. PMID 19654194
- [Background] Papaioannou A, Kennedy CC, Ioannidis G, Sawka A, Hopman WM, Pickard L, Brown JP, Josse RG, Kaiser S, Anastassiades T, Goltzman D, Papadimitropoulos M, Tenenhouse A, Prior JC, Olszynski WP, Adachi JD; CaMos Study Group. The impact of incident fractures on health-related quality of life: 5 years of data from the Canadian Multicentre Osteoporosis Study. Osteoporos Int. 2009 May;20(5):703-14. doi: 10.1007/s00198-008-0743-7. Epub 2008 Sep 19. PMID 18802659
- [Background] Wiktorowicz ME, Goeree R, Papaioannou A, Adachi JD, Papadimitropoulos E. Economic implications of hip fracture: health service use, institutional care and cost in Canada. Osteoporos Int. 2001;12(4):271-8. doi: 10.1007/s001980170116. PMID 11420776
- [Background] Papaioannou A, Morin S, Cheung AM, Atkinson S, Brown JP, Feldman S, Hanley DA, Hodsman A, Jamal SA, Kaiser SM, Kvern B, Siminoski K, Leslie WD; Scientific Advisory Council of Osteoporosis Canada. 2010 clinical practice guidelines for the diagnosis and management of osteoporosis in Canada: summary. CMAJ. 2010 Nov 23;182(17):1864-73. doi: 10.1503/cmaj.100771. Epub 2010 Oct 12. No abstract available. PMID 20940232
- [Background] Martyn-St James M, Carroll S. Meta-analysis of walking for preservation of bone mineral density in postmenopausal women. Bone. 2008 Sep;43(3):521-31. doi: 10.1016/j.bone.2008.05.012. Epub 2008 May 26. PMID 18602880
- [Background] Gillespie LD, Robertson MC, Gillespie WJ, Lamb SE, Gates S, Cumming RG, Rowe BH. Interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD007146. doi: 10.1002/14651858.CD007146.pub2. PMID 19370674
- [Background] Eakin EG, Glasgow RE, Riley KM. Review of primary care-based physical activity intervention studies: effectiveness and implications for practice and future research. J Fam Pract. 2000 Feb;49(2):158-68. PMID 10718694
- [Background] Health Council of Canada 2010. Family Physicians as Gatekeepers.
- [Background] Abramson S, Stein J, Schaufele M, Frates E, Rogan S. Personal exercise habits and counseling practices of primary care physicians: a national survey. Clin J Sport Med. 2000 Jan;10(1):40-8. doi: 10.1097/00042752-200001000-00008. PMID 10695849
- [Background] Yarnall KS, Pollak KI, Ostbye T, Krause KM, Michener JL. Primary care: is there enough time for prevention? Am J Public Health. 2003 Apr;93(4):635-41. doi: 10.2105/ajph.93.4.635. PMID 12660210
- [Background] Petrella RJ, Wight D. An office-based instrument for exercise counseling and prescription in primary care. The Step Test Exercise Prescription (STEP). Arch Fam Med. 2000 Apr;9(4):339-44. doi: 10.1001/archfami.9.4.339. PMID 10776362
- [Background] Nupponen R. What is counseling all about--basics in the counseling of health-related physical activity. Patient Educ Couns. 1998 Apr;33(1 Suppl):S61-7. doi: 10.1016/s0738-3991(98)00010-x. PMID 10889747
- [Background] Ritchie CS, Stetson BA, Bass PF 3rd, Adams KJ. Talking to patients about aerobic exercise for disease prevention: an educational exercise for medical students. Nutr Clin Care. 2002 May-Jun;5(3):103-14. doi: 10.1046/j.1523-5408.2002.00041.x. PMID 12134565
- [Background] Walsh JM, Swangard DM, Davis T, McPhee SJ. Exercise counseling by primary care physicians in the era of managed care. Am J Prev Med. 1999 May;16(4):307-13. doi: 10.1016/s0749-3797(99)00021-5. PMID 10493287
- [Background] Health Canada. Database on the Internet 2011; Available at: http://www.hc-sc.gc.ca/hl-vs/physactiv/index-eng.php. Accessed June 8 2011.
- [Background] Barling NR, Lehmann M. Young men's awareness, attitudes and practice of testicular self-examination: a Health Action Process Approach. Psychol Health Med 1999; 4(3):255-263.
- [Background] Cao D, Xie G. From intention to health behavior: An overview on Health Action Process Approach. Chinese Journal of Clinical Psychology 2010; 18(6):809-812.
- [Background] Chiu C. Testing schwarzer's health action process approach (HAPA) model of health promotion for people with multiple sclerosis: A path analytic approach. University of Wisconsin - Madison; 2009. 217 pp. Available from: UMI Order AAI3384139.:M1: Ph.D.
- [Background] Luszczynska A, Goc G, Scholz U, Kowalska M, Knoll N. Enhancing intentions to attend cervical cancer screening with a stage-matched intervention. Br J Health Psychol. 2011 Feb;16(Pt 1):33-46. doi: 10.1348/135910710X499416. PMID 21226782
- [Background] Schwarzer R, Luszczynska A. How to overcome health-compromising behaviors: The health action process approach. European Psychologist 2008; 13(2):141-151.
- [Background] Williams RJ, Herzog TA, Simmons VN. Risk perception and motivation to quit smoking: a partial test of the Health Action Process Approach. Addict Behav. 2011 Jul;36(7):789-91. doi: 10.1016/j.addbeh.2011.03.003. Epub 2011 Mar 21. PMID 21463920
- [Background] Schwarzer R. Self-efficacy: Thought control of action. Self-efficacy in the adoption and maintenance of health behaviors: Theoretical approaches and a new model. Washington: Hemisphere; 1992. p. 217-243.
- [Background] Luszczynska A, Schwarzer R. Planning and self-efficacy in the adoption and maintenance of breast self-examination: A longitudinal study on self-regulatory cognitions. Psychology and Health 2003; 18:93-108.
- [Background] Renner B, Spivak Y, Kwon S, Schwarzer R. Does age make a difference? Predicting physical activity of South Koreans. Psychol Aging. 2007 Sep;22(3):482-93. doi: 10.1037/0882-7974.22.3.482. PMID 17874949
- [Background] Buman MP, Hekler EB, Haskell WL, Pruitt L, Conway TL, Cain KL, Sallis JF, Saelens BE, Frank LD, King AC. Objective light-intensity physical activity associations with rated health in older adults. Am J Epidemiol. 2010 Nov 15;172(10):1155-65. doi: 10.1093/aje/kwq249. Epub 2010 Sep 15. PMID 20843864
- [Background] Gerdhem P, Dencker M, Ringsberg K, Akesson K. Accelerometer-measured daily physical activity among octogenerians: results and associations to other indices of physical performance and bone density. Eur J Appl Physiol. 2008 Jan;102(2):173-80. doi: 10.1007/s00421-007-0571-z. Epub 2007 Sep 29. PMID 17906874
- [Background] Matthews CE, Ainsworth BE, Thompson RW, Bassett DR Jr. Sources of variance in daily physical activity levels as measured by an accelerometer. Med Sci Sports Exerc. 2002 Aug;34(8):1376-81. doi: 10.1097/00005768-200208000-00021. PMID 12165695
- [Background] Hughes DA. Feasibility, validity and reliability of the Welsh version of the EQ-5D health status questionnaire. Qual Life Res. 2007 Oct;16(8):1419-23. doi: 10.1007/s11136-007-9238-9. Epub 2007 Jul 25. PMID 17653613

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No pre-assignment of participants to groups.
Groups:
- Identify Patients at Risk/Exercise Prescription: The intervention was delivered in two visits and two follow-up phone calls. Physician identifies that the patient is at risk of falls or fractures Visit one: individualized exercise prescription by a physiotherapist.Visit two: motivational interviewing (behavioural counselling) by kinesiologist Phone call 1 and 2: Kinesiologist reviews behavioural components (action planning, coping planning, coping self-efficacy, intentions.
Period: Overall Study
Arm/Group | Identify Patients at Risk/Exercise Prescription
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Identify Patients at Risk/Exercise Prescription: The intervention was delivered in two visits and two follow-up phone calls. Physician identifies that the patient is at risk of falls or fractures Visit one: individualized exercise prescription by a physiotherapist. Visit two: motivational interviewing (behavioural counselling) by kinesiologist Phone call 1 and 2: Kinesiologist reviews behavioural components (action planning, coping planning, coping self-efficacy, intentions.
  Identification of patients at risk, tailored exercise prescription, motivational interviewing, review of behavioural outcomes: The intervention was delivered in two visits and two follow-up phone calls.
Arm/Group | Identify Patients at Risk/Exercise Prescription
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 11
Sedentary [Mean (Standard Deviation); unit: min/day] | 546.2 (274.7)
Low Light Physical Activity [Mean (Standard Deviation); unit: min/day] | 211.3 (100.0)
High Light Physical Activity [Mean (Standard Deviation); unit: min/day] | 32.8 (24.4)
Moderate to Vigorous Physical Activity [Mean (Standard Deviation); unit: min/day] | 24.7 (22.8)
Short Physical Performance Battery [Mean (Standard Deviation); unit: units on a scale] — Short Physical Performance Battery Served as a Functional Assessment at Baseline and Follow-up: 0 (represents worst performance) to 12 (represents best performance).
  units on a scale | 7.91 (3.02)
Timed Up and Go (TUG) [Mean (Standard Deviation); unit: seconds] — Timed Up and Go was a functional assessment taken at baseline and follow-up. A score of more than or equal to 14 seconds has been shown to indicate high risk of falls.
  seconds | 13.95 (6.12)
Coping Planning [Mean (Standard Deviation); unit: units on a scale] — Psychometric questionnaire assessing coping planning was administered at baseline and follow-up. The psychometric questionnaire used a 5 point Likert scale to assess four constructs related to planning behaviour for interference in the participant's exercise routine. The minimum score of 4 represents the least degree of concrete planning for mitigate interference to the participant's exercise routine and the maximal score of 20 indicates a high degree of planning.
  units on a scale | 10.45 (3.93)
Action Planning [Mean (Standard Deviation); unit: units on a scale] — Psychometric questionnaire assessing Action Planning was administered at baseline and follow-up. The psychometric questionnaire used a 5 point likert scale to assess five constructs related to planning behaviour for creating the participant's exercise routine. The minimum score of 5 represents the least degree of concrete planning for the participant's exercise routine and the maximal score of 25 indicates a high degree of planning.
  units on a scale | 16.45 (5.66)
Coping Self-Efficacy [Mean (Standard Deviation); unit: units on a scale] — Psychometric questionnaire assessing Coping Self-Efficacy was administered at baseline and follow-up. The psychometric questionnaire used a 5 point likert scale to assess eight constructs related to self-reported psychological interference in the participant's exercise routine. The minimum score of 8 represents the least amount of self-reported ability to mitigate interference to the participant's exercise routine and the maximal score of 45 indicates a high degree of self-reported resilience .
  units on a scale | 32.55 (6.59)
Intentions [Mean (Standard Deviation); unit: units on a scale] — Psychometric questionnaire assessing Intentions was administered at baseline and follow-up. The psychometric questionnaire used a 5 point likert scale to assess three constructs related to the participant's intentions for exercising over the next 6 weeks. The minimum score of 3 represents the least degree of intention to exercise at the prescribed amount over the next 6 weeks and the maximal score of 15 indicates a high degree of intention to exercise.
  units on a scale | 11.73 (2.20)
EQ-5D-5L (HRQOL) [Mean (Standard Deviation); unit: units on a scale] — The EQ-5D-5L questionnaire will be used to assess health related quality of life at baseline and at six weeks follow-up. The EQ-5D-5L questionnaire is very short and easy to complete making it ideal for a busy clinical setting. It consists of five questions which ask about pain, depression, activities, self-care and mobility. 0 (represents best performance) to 25 (represents worst performance).
  units on a scale | 7.05 (1.19)

OUTCOME MEASURES:

1. Primary Outcome: Physical Activity (Reporting Change in Physical Activity From Baseline to Six-week Follow-up)
Description: The X2-Mini accelerometer (Gulf Coast Data Concepts.,USA) is a three-dimensional sensor that is used to capture the activity levels of an individual. The accelerometer is worn on the hip of the participant for four days. The number of minutes that the individual spends in each exercise intensity category is acquired. Accelerometer thresholds make up four categories of activity: (1) sedentary; (2) low-light; (3) high-light; (4) moderate-vigorous. Activity monitors have been indicated as the most accurate means of measuring physical activity levels.
Time Frame: Baseline, 6 week follow-up
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Identify Patients at Risk/Exercise Prescription
Number analyzed (Participants) | 11
minutes/day | 21.6 (15.8)

2. Primary Outcome: Physical Activity (Self-report) (Reporting Change in Physical Activity From Baseline to Six-week Follow-up)
Description: Participants complete a physical activity log book daily in order to document their completion of the prescribed exercises and list any additional activities that they may have been engaged in. The percentage of prescribed exercises completed are reported (for e.g. if participants completed 2 of 3 prescribed exercise then the reported percentage would be 67%). Mean (SD) are reported.
Time Frame: Baseline, 6 week follow-up
Measure: Mean (Standard Deviation); unit: percentage of completed exercise
Arm/Group | Identify Patients at Risk/Exercise Prescription
Number analyzed (Participants) | 11
percentage of completed exercise | 65.7 (23.2)

3. Secondary Outcome: Behavior Change Outcome: Action Planning
Description: A psychometric questionnaire will assess action planning using a likert scale at baseline and 6 weeks follow-up.
  Action Planning: when, where and how an individual will engage in the recommended exercise. Psychometric questionnaire assessing Action Planning was administered at baseline and follow-up. The psychometric questionnaire used a 5 point likert scale. (0 represents worst performance) to 25 (best performance).
Time Frame: Baseline, 6 week follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Identify Patients at Risk/Exercise Prescription
Number analyzed (Participants) | 11
units on a scale | 21.00 (1.79)

4. Secondary Outcome: Behavior Change Outcome: Coping Planning
Description: A psychometric questionnaire will assess coping planning using a likert scale at baseline and 6 weeks follow-up.
  Coping Planning: assesses an individuals ability to overcome perceived barriers e.g. lack of time, poor weather. Psychometric questionnaire assessing coping planning was administered at baseline and follow-up. The psychometric questionnaire used a 5 point likert scale. (0 represents worst performance) to 20 (best performance).
Time Frame: Baseline, 6 week follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Identify Patients at Risk/Exercise Prescription
Number analyzed (Participants) | 11
units on a scale | 14.55 (1.92)

5. Secondary Outcome: Behavior Change Outcome: Coping Self-Efficacy
Description: A psychometric questionnaire will assess coping self-efficacy using a likert scale at baseline and 6 weeks follow-up.
  Coping Self-Efficacy: assesses an individuals belief in their ability to overcome barriers. Psychometric questionnaire assessing Coping Self-Efficacy was administered at baseline and follow-up. The psychometric questionnaire used a 5 point likert scale. (0 represents worst performance) to 45 (best performance).
Time Frame: Baseline, 6 week follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Identify Patients at Risk/Exercise Prescription
Number analyzed (Participants) | 11
units on a scale | 34.45 (4.11)

6. Secondary Outcome: Behavior Change Outcome: Intentions
Description: A psychometric questionnaire will assess intentions using a likert scale at baseline and 6 weeks follow-up.
  Intentions: assesses an individuals intention to engage in recommended exercises. Psychometric questionnaire assessing Intentions was administered at baseline and follow-up. The psychometric questionnaire used a 5 point likert scale. (0 represents worst performance) to 15 (best performance).
Time Frame: Baseline, 6 week follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Identify Patients at Risk/Exercise Prescription
Number analyzed (Participants) | 11
units on a scale | 12.0 (1.61)

7. Secondary Outcome: Health Related Quality of Life (HRQOL)
Description: The EQ-5D-5L questionnaire will be used to assess health related quality of life at baseline and at six weeks follow-up. The EQ-5D-5L questionnaire is very short and easy to complete making it ideal for a busy clinical setting. It consists of five questions which ask about pain, depression, activities, self-care and mobility. 0 (represents best performance) to 25 (represents worst performance).
Time Frame: Baseline, 6 week follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Identify Patients at Risk/Exercise Prescription
Number analyzed (Participants) | 11
units on a scale | 8.0 (1.0)
Statistical Analysis 1: Comparison: Identify Patients at Risk/Exercise Prescription; Test type: Other; p < 0.05, Wilcoxon (Mann-Whitney) — <0.05 (threshold for significance)

ADVERSE EVENTS:
Arm/Group | Identify Patients at Risk/Exercise Prescription
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

LIMITATIONS AND CAVEATS:
Small sample size and short study duration. Use of accelerometers to objectively capture physical activity (not all activity is captured by the accelerometers) and use of self-report physical activity logs. Possible self motivated participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No